CLINICAL TRIAL: NCT02947698
Title: Effect of Weekend Admission on Mortality Associated With Severe Acute Kidney Injury in England: a Propensity Score Matched, Population-based Study
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Nitin Kolhe, Consultant Nephrologist, University Hospitals of Derby and Burton NHS Foundation Trust
Other Study IDs: 1.4
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Acute Kidney Injury; Outcome, Fatal
Keywords: acute kidney injury; weekend admission; mortality
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute kidney injury patients admitted on weekday: All patients with acute kidney injury requiring dialysis admitted on week day (Monday to Friday) between 1st April 2003 and 31st March 2015
- Acute kidney injury patients admitted on weekend: All patients with acute kidney injury requiring dialysis admitted on weekend (Saturday or Sunday) between 1st April 2003 and 31st March 2015

SUMMARY:
Increased in-hospital mortality associated with weekend admission has been reported for many acute conditions, but no study has investigated "weekend effect" for acute kidney injury requiring dialysis (AKI-D). In this study, the investigators compared mortality in AKI-D patients admitted on weekday versus weekend and assessed factors associated with increased mortality.

DETAILED DESCRIPTION:
Several studies have reported an unwanted adverse effect of weekend admission on mortality in certain acute medical conditions. Though the reason for this variation could be illness severity, some studies have hypothesized that this could be due to variation in care provided over weekends when services are a minimum. The increased mortality over weekends for certain conditions in the National Health Service (NHS) in England has led to an intense debate on reconfiguring the health service. Little is known about the impact of the weekend effect on severe acute kidney requiring dialysis (AKI-D) in England, the incidence of which has increased more than 12-foldover the past 15 years. Most nephrology departments in England provide continuous consultant cover over weekends and have the capacity to perform emergency dialysis as needed over weekends suggesting that a weekend effect is less likely to occur. Patients admitted over the weekend may present in three ways - with severe AKI requiring dialysis over the weekend, with AKI and requiring dialysis on a subsequent weekday or with no AKI, but develop AKI-D during the in-patient stay over next few days. Some studies have reported that patients starting dialysis on Sunday or a diagnosis of severe AKI over weekend, does not affect mortality, while others have reported increased mortality for AKI in all sizes of hospital over weekend. One explanation for this observation is that necessary dialysis therapy may not be initiated on a weekend as a result of limitations in physician or nurse staffing or device availability. However, bias can be created by single center studies as it is well recognized that the epidemiology of AKI-D shows considerable regional variation and this may be true for all days of the week. It can also be speculated that patients admitted on weekends may not receive optimal care resulting in development of new AKI or progression of AKI to AKI-D resulting in excess mortality.

With this background, the investigators wanted to investigate whether a weekend effect on mortality exists for AKI-D patients in England. The investigators hypothesized that patients admitted over weekend would have increased mortality irrespective of demographic features and clinical characteristics. They also hypothesized that the effect on mortality would be more pronounced in centers with no on-site nephrology services.

ELIGIBILITY:
Inclusion Criteria:

1. AKI cases identified by using validated International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) codes of N17 in any diagnoses codes.
2. AKI cases requiring dialysis (AKI-D) were identified by OPCS code of X40.3 for hemodialysis or X40.4 for hemofiltration in any of the 24 procedures.

Exclusion Criteria:

1. Patients' with ICD10 codes N18.5 and N18.6 for chronic kidney disease stage five (CKD-5) and end stage renal disease (ESRD) respectively will be excluded.
2. Patients with OPCS-4 codes for arteriovenous fistula (L74.2) or arteriovenous shunt (L74.3) during the inpatient admission will be excluded.

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 2003-2015 data from the Hospital Episode Statistics (HES) database containing details of all admissions at National Health Service (NHS) hospitals in England will be used to extract all AKI-D patients
Sampling Method: Probability Sample
Enrollment: 53878 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality for weekend and weekday AKI-D admissions | 60-day

SECONDARY OUTCOMES:
Effect of in-center nephrology services on weekdays and weekend mortality of AKI-D admissions | 60-day
Effect of deprivation on weekdays and weekend mortality of AKI-D admissions | 60-day
  The Index of Multiple Deprivation is the official measure of relative deprivation (for neighborhoods) in England. The Index of Multiple Deprivation ranks every small area in England from one (most deprived area) to 32,844 (least deprived area) and deciles are calculated dividing the ranking into 10 equal groups

CONTACTS AND LOCATIONS:
Overall Officials: Nitin V Kolhe, MD, Principal Investigator — Derby Hospital NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
The data is anonymised and freely available from HSCIC